CLINICAL TRIAL: NCT02656537
Title: EnSite™ HD Grid Catheter Mapping System for Advanced High Density Three-Dimensional Mapping in Non-Paroxysmal Atrial Fibrillation and Atrial Tachycardia
Brief Title: EnSite™ HD Grid Catheter AF/AT Mapping Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CRD772
Record Dates: First submitted 2015-11-16; First posted 2016-01-15 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Non-paroxysmal Atrial Fibrillation; Left Atrial Tachycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EnSite™ HD Grid Catheter AF/AT Mapping (Experimental)
  Interventions: Device: EnSite™ HD Grid Catheter mapping system

INTERVENTIONS:
Device: EnSite™ HD Grid Catheter mapping system

SUMMARY:
In this clinical investigation, the safety, feasibility and performance of the novel EnSite™ HD Grid Catheter mapping system for advanced high-density three-dimensional mapping will be studied in patients undergoing catheter ablation procedures for the treatment of non-paroxysmal atrial fibrillation (AF) or left atrial tachycardia (AT).

DETAILED DESCRIPTION:
Catheter ablation for non-paroxysmal AF is more complex as triggers, if present at all, are not immediately apparent, but the abnormal atrial substrates are the likely predominant mechanisms. Additional catheter ablation strategies targeting for atrial substrate modification have been introduced. The common strategies involve either application of empirical linear lesion sets in the atrial areas or ablation of atrial areas with complex fractionated atrial electrograms in addition to pulmonary vein isolation. Nevertheless, the corresponding success rates in long-term sinus rhythm maintenance are modest.

Non-paroxysmal AF and left AT are characterized by fast and regular atrial activities, complex fractionated atrial electrograms, consistent direction of wave front propagation, and low peak-to-peak voltage. Advanced high-density three-dimensional catheter mapping strategies to target the evaluation of these characteristics and mechanisms responsible for the AF and left AT, identification of atrial areas with low peak-to-peak voltages and determination of the "critical" atrial targets for catheter ablation during the procedures would be essential.

In this clinical investigation, the safety, feasibility and performance of the novel EnSite™ HD Grid Catheter mapping system for advanced high-density three-dimensional mapping will be studied in patients undergoing catheter ablation procedures for the treatment of non-paroxysmal AF or left AT.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of non-paroxysmal atrial fibrillation (AF) or left atrial tachycardia (AT) referred for catheter ablation
2. Age of 18 years of age or older at time of Enrollment
3. On continuous anticoagulation (INR 2-3) for >4 weeks prior to the ablation
4. Able and willing to provide written informed consent to participate in this clinical investigation

Exclusion Criteria:

1. Secondary atrial fibrillation (AF)
2. Presence of a prosthetic valve(s) or hemodynamically significant valvular heart disease as determined by Study Investigator
3. Active systemic infection (e.g. sepsis)
4. Presence of left atrial thrombus (i.e., positive TEE) or myxoma, or interatrial baffle or patch via the transseptal approach
5. Contraindication to systemic anticoagulation (i.e., heparin, warfarin, or a direct thrombin inhibitor)
6. History of cerebrovascular accidents (Stroke, TIA)
7. Previous myocardial infarction, unstable angina pectoris or coronary artery by-pass <180 days at Enrollment or cardiovascular intervention expected in the 180 days post-Enrollment
8. Left atrial size >55mm
9. NYHA (New York Heart Association Classification) functional class III or IV heart failure
10. Left ventricular ejection fraction <35%
11. Uncontrolled Hyperthyroidism
12. Pregnant or of childbearing potential and not using adequate contraceptive methods or nursing
13. Participating in another clinical investigation that may confound the results of this clinical investigation
14. Life expectancy less than 12 months, as determined by Study Investigator
15. Severe clinical condition (e.g. active carcinoma) that, in the opinion of the Study Investigator, excludes the participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events associated with the use of the EnSite™ HD (High-Density)Grid Catheter mapping system. | Within 48 hours from Procedure
  To evaluate the safety of the novel EnSite™ HD Grid Catheter mapping system by collecting intra- and post-Procedure (within 48 hours from Procedure) adverse events.
Number of subjects with the electrophysiological characteristics of non-paroxysmal AF and left AT pre-catheter ablation studied using the EnSite™ HD Grid Catheter mapping system. | During Procedure
  To identify and study the electrophysiological characteristics of non-paroxysmal AF and left AT pre-catheter ablation using a novel EnSite™ HD Grid Catheter mapping system.
Catheter performance during the mapping portion of the procedure | During Procedure
  To assess the HD Grid Catheter mapping system for acceptable geometry creation, map repeatability and electrogram signal quality.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Pappone, MD, PhD, Principal Investigator — San Donato Hospital, Italy
Locations (7):
- Australia (3):
  - Royal Adelaide Hospital, Adelaide
  - Ashford Hospital, Ashford
  - Royal Melbourne Hospital, Parkville
- Hôpital du Haut Lévêque, Pessac, France
- Herzzentrum Dresden GmbH Universitatsklinik, Dresden, Germany
- Queen Mary Hospital, Hong Kong, Hong Kong
- San Donato Hospital, Milan, Italy